CLINICAL TRIAL: NCT05424835
Title: A Phase III, Multicenter, Randomized, Open-Label, Parallel Controlled Study of SHR-A1811 Versus Pyrotinib in Combination With Capecitabine for HER2-Positive, Unresectable and/or Metastatic Breast Cancer Subjects Previously Treated With Trastuzumab and Taxane
Brief Title: A Trial of SHR-A1811versus Pyrotinib in Combination With Capecitabine in HER2-Positive, Unresectable and/or Metastatic Breast Cancer Subjects Previously Treated With Trastuzumab and Taxane
Status: Active, not recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Jiangsu HengRui Medicine Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: SHR-A1811-III-301
Record Dates: First submitted 2022-06-15; First posted 2022-06-21 (Actual); Last update posted 2025-08-22 (Actual); Status verified 2024-09

CONDITIONS: HER2-Positive, Unresectable and/or Metastatic Breast Cancer Subjects Previously Treated With Trastuzumab and Taxane
MeSH Terms: interventions — pyrotinib; Capecitabine

STUDY DESIGN:
Intervention Model Description: SHR-A1811 compared with Pyrotinib in combination with Capecitabine
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Treatment group A (Experimental): SHR-A1811 4.8mg/kg
  Interventions: Drug: SHR-A1811
- Treatment group B (Active Comparator): Pyrotinib in combination with Capecitabine.
  Interventions: Drug: Pyrotinib in combination with Capecitabine.
- Treatment group C (Experimental): SHR-A1811 6.4mg/kg
  Interventions: Drug: SHR-A1811
- Treatment group D (Active Comparator): Pyrotinib in combination with Capecitabine.
  Interventions: Drug: Pyrotinib in combination with Capecitabine.

INTERVENTIONS:
Drug: SHR-A1811 — SHR-A1811 4.8mg/kg
  Arms: Treatment group A
Drug: Pyrotinib in combination with Capecitabine. — Pyrotinib in combination with Capecitabine.
  Arms: Treatment group B; Treatment group D
Drug: SHR-A1811 — SHR-A1811 6.4mg/kg
  Arms: Treatment group C

SUMMARY:
The study is being conducted to evaluate whether the efficacy of SHR-A1811 is better than Pyrotinib in combination with Capecitabine in HER2-Positive, Unresectable and/or Metastatic Breast Cancer Subjects Previously Treated With Trastuzumab and Taxane.

ELIGIBILITY:
Inclusion Criteria:

1. Able and willing to provide a written informed consent;
2. Unresectable or metastatic HER2 positive breast cancer previously treated with Trastuzumab and Taxane in recurrence and metastasis stage;
3. Documented disease progression;
4. Eastern Cooperative Oncology Group (ECOG) performance status of 0 or 1;
5. Life expectancy ≥ 12 weeks.
6. Subject has measurable disease based on RECIST v1.1;
7. Important organ function can meet the criteria (no blood component and cell growth factor treatment within 14 days before the first study drug administration)
8. Pregnancy and Contraception:

   * Women of childbearing potential (WOCBP) must agree to use highly effective contraceptive measures and not to lactate from screening until 7 months after receiving the last treatment.
   * Women of childbearing potential (WOCBP) must have a negative serum pregnancy test within 7 days prior to the first study drug administration.

Exclusion Criteria:

1. Subjects with other malignant tumors in the past 5 years (except for the cured skin basal cell carcinoma and cervical carcinoma in situ).
2. There is a third interstitial effusion (e.g., massive ascites, pleural effusion, pericardial effusion) that cannot be controlled by drainage or other methods.
3. Inability to swallow, chronic diarrhea, intestinal obstruction, or other factors that affect drug administration and absorption.
4. Received mitomycin C and nitrosoureas chemotherapy within 6 weeks before the first study drug administration.
5. Any surgery (eg., major surgery for cancer), radiotherapy, chemotherapy, immunotherapy or molecular targeted therapy, biotherapy or other drug clinical trial within 4 weeks; received endocrine therapy within 2 weeks before the first study drug administration.
6. Any concurrent use of immunosuppressant or systemic corticosteroid treatment to achieve immunosuppression purpose (dose of > 10mg/day prednisone or equivalent), and still in use within 2 weeks before the first study drug administration.
7. History of autoimmune disease with the possibility of recurrence or active autoimmune disease; subjects with skin diseases without systematic treatment such as vitiligo, psoriasis, alopecia, or controlled type I diabetes treated with insulin can be included; asthma completely relieved in childhood without any intervention in adult can be included, subjects that requires medical intervention with bronchodilators for asthma cannot be included).
8. History of immunodeficiency including seropositivity for human immunodeficiency virus (HIV) or other acquired or congenital immune-deficient disease, or organ transplantation.
9. Cardiac disease including myocardial infarction within a minimum 6 months before the first study drug administration, severe or unstable angina, symptomatic congestive heart failure (New York Heart Association [NYHA] classes ≥II), or clinically significant supraventricular or ventricular cardiac arrhythmia requiring treatment/intervention.
10. Subjects with known or suspected interstitiallung disease;
11. Active hepatitis B (HBsAg positive and HBV DNA ≥ 500 IU / ml), hepatitis C (hepatitis C antibody positive and HCV RNA higher than the detection limit of the analytical method), hepatic cirrhosis, or severe infections requiring antibiotic, antiviral or antifungal control.
12. Unresolved toxicities from previous anticancer therapy, defined as toxicities (other than alopecia) not yet resolved to NCI CTCAE v5.0 Grade ≤1 at baseline. Subjects with chronic Grade 2 toxicities may be eligible at the discretion of the investigator and discussion with sponsor.
13. Known history of severe allergy to study drug or its components, or allergy to humanized monoclonal antibody products (such as trastuzumab, pertuzumab, etc.).
14. The presence of other serious physical or mental disorders or abnormalities in laboratory tests that may increase the risk of study participation or interfere with study results, as well as patients deemed unsuitable for study participation by the investigator.

Ages: 18 Years to 75 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 381 (Actual)
Dates: Start 2022-08-04 (Actual); Primary Completion 2026-12-31 (Estimated); Study Completion 2027-12-31 (Estimated)

PRIMARY OUTCOMES:
PFS（BIRC assessment）between SHR-A1811 4.8mg/kg Q3W and Pyrotinib in combination with Capecitabine. | 6 weeks after the first study drug administration，about 2 years.

SECONDARY OUTCOMES:
PFS（INV assessment）between SHR-A1811 4.8mg/kg Q3W and Pyrotinib in combination with Capecitabine | 6 weeks after the first study drug administration，about 2 years.
ORR between SHR-A1811 4.8mg/kg Q3W and Pyrotinib in combination with Capecitabine； | about 2 years.
DoR between SHR-A1811 4.8mg/kg Q3W and Pyrotinib in combination with Capecitabine； | about 2 years.
OS between SHR-A1811 4.8mg/kg Q3W and Pyrotinib in combination with Capecitabine； | about 4 years.
PFS（BIRC assessment）between SHR-A1811 6.4mg/kg Q3W and Pyrotinib in combination with Capecitabine； | 6 weeks after the first study drug administration，about 2 years.
PFS（INV assessment）between SHR-A1811 6.4mg/kg Q3W and Pyrotinib in combination with Capecitabine； | 6 weeks after the first study drug administration，about 2 years.
ORR between SHR-A1811 6.4mg/kg Q3W and Pyrotinib in combination with Capecitabine； | about 2 years.
DoR between SHR-A1811 6.4mg/kg Q3W and Pyrotinib in combination with Capecitabine； | about 2 years.
OS between SHR-A1811 6.4mg/kg Q3W and Pyrotinib in combination with Capecitabine； | about 4 years.
AE | about 2 years.

CONTACTS AND LOCATIONS:
Locations (1):
- Sun Yat-Sen Memorial Hospital, Sun Yat-Sen University, Guangzhou, Guangdong, China

IPD SHARING:
Plan to Share IPD: Undecided